CLINICAL TRIAL: NCT06980571
Title: Randomised Prospective Study of CUSA Versus Radiofrequency Ablation Technique in Liver Resections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P3/04/Q0605/31
Record Dates: First submitted 2009-01-27; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Liver Disease
Keywords: liver resection; blood loss; resection technique; CUSA; radiofrequency ablation; health economics; benign and malignant liver disease
MeSH Terms: conditions — Liver Diseases; Hemorrhage | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequency ablation (Active Comparator): 50 patients randomised to radiofrequency ablation technique of liver resection
  Interventions: Device: radiofrequency ablation
- CUSA (No Intervention): 50 patients having liver resection randomised to CUSA

INTERVENTIONS:
Device: radiofrequency ablation — FDA approved intervention being compared with gold standard (most common intervention)
  Arms: Radiofrequency ablation

SUMMARY:
The purpose of this study is to determine whether a particular method of operating on the liver is superior to the "gold" standard commonest technique. CUSA (ultrasonic agitation) will be compared to the newer heat coagulation technique (radiofrequency ablation) and comparisons of blood loss, transfusion requirements, complication rates, hospital stay, effect on liver function, health economics and death rate will be made. The groups will be assessed for comparability in terms of underlying disease, resection type, underlying concurrent illnesses, sex, age, background liver disease. Standardisations of the rest of the operation will be carried out including anaesthetic technique and fluid requirements will be assessed by oesophageal Doppler. 100 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* any adult patient listed for liver resection giving informed consent

Exclusion Criteria:

* children, non-consent and diminished responsibility

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-06; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Blood loss per cm squared of liver parenchyma cut through | operation date until three months from discharge

SECONDARY OUTCOMES:
mortality | inpatient and thirty day mortality
  incidence of post-operative complications measured over a thirty day period

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Hutchins, MB BS MS FRCS, Principal Investigator — Royal London Hospital
Locations (1):
- Royal London Hospital, London, United Kingdom